CLINICAL TRIAL: NCT02435381
Title: Carisbamate as a Potential Treatment for Alcohol Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Christopher Verrico, Assistant Professor, Psychiatry Research, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-30334
Record Dates: First submitted 2013-09-07; First posted 2015-05-06 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Alcohol Dependence; Alcohol Abuse; Substance Abuse
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo from days 2- 4.
  Interventions: Drug: Placebo
- Carisbamate (Active Comparator): Participants will receive carisbamate 600mg qd from days 2- 4.
  Interventions: Drug: Carisbamate

INTERVENTIONS:
Drug: Carisbamate — 600mg Orally on days 2-4
  Other Names: YKP 509
  Arms: Carisbamate
Drug: Placebo — Placebo treatment only
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of treatment with carisbamate compared to treatment with placebo, on alcohol-induced stimulant and subjective effects in non-treatment seeking alcohol-dependent human volunteers.

DETAILED DESCRIPTION:
This within-subjects placebo-controlled experimental protocol will assess the effects of carisbamate (600mg qd) on the positive subjective effects of alcohol in non-treatment-seeking alcohol-dependent volunteers. Participants will receive study drug (carisbamate or placebo) from days 2- 4. On day 4, study drug will be followed by alcohol (0.8g/kg; 16% by volume) and a placebo beverage (1% by volume as a mask), both separated by 2 hours. Physiologic, subjective effects and BAL will be obtained after the alcohol challenges. Participants will be discharged on day 4 and asked to return a week later to repeat the study under the alternate study drug condition (active carisbamate vs. placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Be an English-speaking volunteer who is not seeking treatment at the time of the study
2. Be between 18-55 years of age
3. Meet DSM-IV TR criteria for alcohol abuse; participants may or may not meet criteria for nicotine dependence. Nicotine dependence is allowed but not required because most alcohol users smoke cigarettes.
4. Have a self-reported history of using alcohol.
5. Have vital signs as follows: resting pulse must be < 90 bpm and the blood pressure must be < 150 mmHg systolic and < 90 mmHg diastolic.
6. Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions:

   * liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) within normal limits
7. Have a baseline EKG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant arrhythmias
8. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.

Exclusion Criteria:

1. Meet DSM IV TR criteria for dependence on drugs other than alcohol or nicotine.
2. Have any history or evidence suggestive of seizure disorder or brain injury
3. Have any previous medically adverse reaction to alcohol, including loss of consciousness, chest pain, or epileptic seizure
4. Have neurological or psychiatric disorders, such as:

   * psychosis, bipolar illness or major depression as assessed by SCID
   * organic brain disease or dementia assessed by clinical interview
   * history of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult
   * history of suicide attempts within the past year and/or current suicidal ideation/plan
5. Have evidence of clinically significant heart disease or hypertension, as determined by the PI
6. Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
7. Have symptomatic HIV or are taking antiretroviral medication
8. Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, upon hospital admission, and at the end of study participation
9. Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.
10. Currently seeking help for alcohol dependence.
11. Subjects with or prone to clinically significant alcohol withdrawal.
12. More than thirty days of abstinence from alcohol in the ninety days prior to enrollment.
13. A history of major alcohol-related medical complications requiring hospitalization (i.e. pancreatitis).
14. Contraindication(s) to take the study medication such as renal or hepatic impairment, nephrolithiasis, congenital metabolic disorders or history of seizures. Moderate-to-severe renal impairment defined as creatinine clearance less than 30 mL/min.
15. Use of inhibitors/substrates for renal cationic transporters, or medications contraindicated with ethanol.
16. A history of violence or aggression, assessed as part of the clinical interview at screening visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Newton, M.D, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a crossover design, double-blind, placebo controlled, 8 week clinical trail.
Groups:
- Placebo First, Then Carisbamate: Participants received placebo from days 2- 4. Participants were discharged on day 4 and asked to return a week later to repeat the study under the alternate study drug condition (active carisbamate)
- Carisbamate First, Then Placebo: Participants received carisbamate from days 2- 4. Participants were discharged on day 4 and asked to return a week later to repeat the study under the alternate study drug condition (placebo)
Period: Overall Study
Arm/Group | Placebo First, Then Carisbamate | Carisbamate First, Then Placebo
Started | 5 | 6
Completed | 3 | 5
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Carisbamate: This within-subjects study included two treatment arms (placebo and carisbamate); 8 subjects completed both study arms.
  Participants received placebo on study days 2- 4. Participants were discharged on day 4 and asked to return a week later to repeat the study procedures under the alternate study drug condition (active carisbamate)
  Placebo: 0mg orally on days 2-4 Carisbamate: 600mg orally on days 2-4
Arm/Group | Placebo/Carisbamate
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
U.S. Veteran [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Biphasic Alcohol Effects Scale (BAES) Scores
Description: The Biphasic Alcohol Effects Scale (BAES) is a self-report, unipolar adjective rating scale that is designed to measure both stimulant and sedative effects of alcohol. The BAES consists of 14 items that are rated on a eleven-point scale. The Sedation and Stimulation subscales are calculated by summing the following items (for the 14-point scale): Stimulation: = BAES3 + BAES4 + BAES5 + BAES11 + BAES12 + BAES13 +BAES14/ Sedation: = BAES1 + BAES2 + BAES6 + BAES7 + BAES8 + BAES9 + BAES10. Individuals are instructed to rate the extent to which drinking alcohol has produced these feelings in you at the present time from 0 (not at all) to 10 (extremely). Higher scores on the Sedative Subscale represent extreme sedation (0 not at all sedated - 70 extremely sedated). Higher scores on the Stimulant Subscale represent extreme stimulation (0 not at all stimulated - 70 extremely stimulated). Scale scores are calculated as the sum of respective stimulant and sedative effects items.
Time Frame: 15, 30 and 60 minutes after consumption of placebo (1% alcohol by volume) and alcohol (0.8g/kg; 16% by volume) beverages, stimulant ratings
Population: This within-subjects study included 2 treatment arms (placebo & carisbamate), during both arms subjects completed study procedures twice, once after consuming placebo (1% alcohol by volume) and once after consuming alcohol (0.8g/kg; 16% by volume). The data here represent the means, following consumption of alcohol and placebo beverage, for the 8 subjects that completed both study arms.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo + Alcohol Beverage; Placebo + Placebo Beverage: Participants will receive placebo from days 2- 4.
  Placebo: Placebo treatment only
- Carisbamate + Alcohol Beverage; Carisbamate + Placebo Beverage: Participants will receive carisbamate 600mg qd from days 2- 4.
  Carisbamate: 600mg Orally on days 2-4
Arm/Group | Placebo + Alcohol Beverage | Carisbamate + Alcohol Beverage | Placebo + Placebo Beverage | Carisbamate + Placebo Beverage
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  'BAES Stimulant Subscale' +15 minutes after alcohol and placebo beverage consumption | 27.5 (5.8) | 32.4 (4.1) | 23.0 (6.9) | 21.1 (5.2)
  'BAES Stimulant Subscale' +30 minutes after alcohol and placebo beverage consumption | 34.4 (4.5) | 32.5 (4.1) | 26.0 (6.6) | 18.5 (4.8)
  'BAES Stimulant Subscale' +60 minutes after alcohol and placebo beverage consumption | 24.8 (6.2) | 29.0 (7.2) | 20.6 (6.0) | 20.1 (5.1)
  'BAES Sedative Subscale' +15 minutes after alcohol and placebo beverage consumption | 16.9 (4.9) | 16.8 (5.1) | 4.9 (2.6) | 11.8 (5.7)
  'BAES Sedative Subscale' +30 minutes after alcohol and placebo beverage consumption | 20.0 (6.1) | 20.4 (6.5) | 7.6 (3.8) | 8.8 (5.3)
  'BAES Sedative Subscale' +60 minutes after alcohol and placebo beverage consumption | 16.8 (5.9) | 20.1 (7.1) | 5.3 (3.0) | 9.5 (5.3)

2. Primary Outcome: Mean Alcohol Urge Questionnaire (AUQ) Scores
Description: The Alcohol Urge Questionnaire (AUQ) consists of eight statements about the respondent's feelings and thoughts about drinking as they are completing the questionnaire (i.e., right now). Drinking refers to various types of alcohol, including beer, wine and liquor. The respondent is asked to respond to each statement about alcohol craving via a 7-item Likert scale ranging from "0-strongly disagree" to "6- strongly agree." Item scores were averaged and the total score also ranges from 0-6.
Time Frame: 15, 30 and 60 minutes after consumption of placebo (1% alcohol by volume) and alcohol (0.8g/kg; 16% by volume) beverages.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo + Alcohol Beverage: Participants will receive placebo from days 2- 4. Participants were discharged on day 4 and asked to return a week later to repeat the study under the alternate study drug condition (active carisbamate)
  Placebo: Placebo treatment only
- Carisbamate + Alcohol Beverage: Participants will receive carisbamate 600mg qd from days 2- 4. Participants were discharged on day 4 and asked to return a week later to repeat the study under the alternate study drug condition ( placebo).
  Carisbamate: 600mg Orally on days 2-4
Arm/Group | Placebo + Alcohol Beverage | Carisbamate + Alcohol Beverage | Placebo + Placebo Beverage | Carisbamate + Placebo Beverage
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  'AUQ' +15 minutes after alcohol and placebo beverage consumption | 3.3 (0.4) | 3.5 (0.5) | 3.1 (0.4) | 3.3 (0.5)
  'AUQ' +30 minutes after alcohol and placebo beverage consumption | 3.7 (0.4) | 3.9 (0.5) | 2.9 (0.5) | 3.4 (0.5)
  'AUQ' +60 minutes after alcohol and placebo beverage consumption | 2.8 (0.5) | 3.4 (0.6) | 3.1 (0.5) | 2.8 (0.5)

3. Primary Outcome: Mean Positive and Negative Affect Schedule (PANAS) Scores
Description: The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much). Range between 10 and 50 points. Higher positive affect scores indicated a better outcome, while lower negative affect scores indicated a better outcome.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Alcohol Beverage | Carisbamate + Alcohol Beverage | Placebo + Placebo Beverage | Carisbamate + Placebo Beverage
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  'PANAS, Positive' +15 minutes after alcohol and placebo beverage consumption | 28.1 (3.4) | 27.5 (3.0) | 27.5 (3.3) | 26.6 (3.4)
  'PANAS, Positive' +30 minutes after alcohol and placebo beverage consumption | 28.4 (3.2) | 29.3 (3.5) | 27.9 (2.8) | 26.6 (3.0)
  'PANAS, Positive' +60 minutes after alcohol and placebo beverage consumption | 29.0 (2.2) | 27.6 (2.9) | 29.3 (2.9) | 28.5 (2.8)
  'PANAS, Negative' +15 minutes after alcohol and placebo beverage consumption | 13.9 (2.0) | 13.0 (1.7) | 12.0 (1.2) | 13.6 (1.8)
  'PANAS, Negative' +30 minutes after alcohol and placebo beverage consumption | 13.3 (2.0) | 13.9 (1.6) | 13.0 (2.5) | 14.3 (1.8)
  'PANAS, Negative' +60 minutes after alcohol and placebo beverage consumption | 13.1 (2.5) | 14.1 (2.6) | 12.9 (2.2) | 15.8 (2.5)

4. Primary Outcome: MEAN DRUG EFFECTS QUESTIONNAIRE (DEQ) SCORES
Description: Self-reported subjective drug effects questionnaire evaluated whether a respondent was currently affected by doses of alcohol. Participants completed VAS at regular intervals after ingesting active alcohol (0.8g/kg; 16% by volume) or placebo (1% by volume as a mask). The questionnaire assessed the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", and "Want More". The "Feel Drug", "Feel High", "Like Drug", "Dislike Drug", and "Want More" subscales are reported.Each item is rated on a 100-point scale of 1 (not at all) to 100 (extremely). 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Alcohol Beverage | Carisbamate + Alcohol Beverage | Placebo + Placebo Beverage | Carisbamate + Placebo Beverage
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  'FEEL' +15 minutes after alcohol and placebo beverage consumption | 32.4 (12.3) | 53.2 (14.4) | 14.0 (12.3) | 23.6 (14.6)
  'FEEL' +30 minutes after alcohol and placebo beverage consumption | 39.4 (11.6) | 53.5 (14.2) | 10.9 (9.3) | 16.8 (10.4)
  'FEEL' +60 minutes after alcohol and placebo beverage consumption | 43.6 (12.8) | 42.6 (13.5) | 11.4 (10.1) | 16.5 (11.0)
  'LIKE' +15 minutes after alcohol and placebo beverage consumption | 46.5 (13.5) | 54.0 (13.6) | 23.1 (10.2) | 33.4 (14.5)
  'LIKE' +30 minutes after alcohol and placebo beverage consumption | 54.8 (13.2) | 47.8 (15.2) | 27.4 (13.4) | 17.6 (10.6)
  'LIKE' +60 minutes after alcohol and placebo beverage consumption | 37.9 (13.1) | 33.8 (11.8) | 18.6 (11.0) | 24.4 (12.0)
  'DISLIKE' +15 minutes after alcohol and placebo beverage consumption | 14.8 (8.9) | 22.8 (14.1) | 18.9 (12.3) | 24.1 (12.6)
  'DISLIKE' +30 minutes after alcohol and placebo beverage consumption | 13.9 (7.6) | 21.9 (14.3) | 22.4 (14.1) | 15.6 (12.2)
  'DISLIKE' +60 minutes after alcohol and placebo beverage consumption | 16.1 (12.1) | 18.0 (11.0) | 22.3 (14.1) | 35.3 (14.2)
  'HIGH' +15 minutes after alcohol and placebo beverage consumption | 35.6 (10.9) | 53.8 (14.4) | 8.8 (6.7) | 31.6 (15.7)
  'HIGH' +30 minutes after alcohol and placebo beverage consumption | 43.0 (10.6) | 52.1 (13.6) | 10.3 (8.6) | 13.8 (10.4)
  'HIGH' +60 minutes after alcohol and placebo beverage consumption | 37.9 (13.5) | 46.9 (14.3) | 1.9 (1.3) | 10.1 (10.1)
  'WANT MORE' +15 minutes after alcohol and placebo beverage consumption | 44.3 (14.3) | 50.5 (14.0) | 24.1 (12.3) | 28.9 (14.7)
  'WANT MORE' +30 minutes after alcohol and placebo beverage consumption | 46.5 (14.5) | 56.3 (15.0) | 30.1 (12.4) | 23.4 (11.7)
  'WANT MORE' +60 minutes after alcohol and placebo beverage consumption | 37.6 (12.6) | 50.0 (15.7) | 28.3 (11.9) | 15.4 (10.2)

5. Secondary Outcome: Physiologic Effects of Carisbamate: Mean Systolic and Diastolic Blood Pressure
Description: systolic and diastolic blood pressure will be monitored after consuming carisbamate and alcohol
Time Frame: 15, 30 and 60 minutes after alcohol (0.8 mg/kg;16% by volume) consumption
Population: This within-subjects study included 2 treatment arms (placebo & carisbamate), during both arms subjects completed study procedures twice, once after consuming placebo and once after consuming alcohol (0.8g/kg; 16% by volume). The data here represent the means, following consumption of alcohol only, for the 8 subjects that completed both study arms.
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Placebo: Participants will receive placebo from days 2- 4. Participants were discharged on day 4 and asked to return a week later to repeat the study under the alternate study drug condition (active carisbamate)
  Placebo: Placebo treatment only
- Carisbamate: Participants will receive carisbamate 600mg qd from days 2- 4. Participants were discharged on day 4 and asked to return a week later to repeat the study under the alternate study drug condition ( placebo).
  Carisbamate: 600mg Orally on days 2-4
Arm/Group | Placebo | Carisbamate
Number analyzed (Participants) | 8 | 8
mm Hg
  'Systolic BP' + 15 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 149.4 (7.1) | 140.1 (7.6)
  'Systolic BP' + 30 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 145.0 (8.0) | 137.3 (5.8)
  'Systolic BP' + 60 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 140.8 (10.5) | 134.0 (8.5)
  'Diastolic BP' + 15 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 89.6 (4.4) | 87.4 (3.0)
  'Diastolic BP' + 30 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 84.4 (4.2) | 84.3 (2.5)
  'Diastolic BP' + 60 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 81.6 (3.9) | 79.6 (3.5)

6. Secondary Outcome: Physiologic Effects of Carisbamate: Mean Heart Rate
Description: pulse will be monitored after consuming carisbamate and alcohol
Time Frame: 15, 30 and 60 minutes after alcohol (0.8 mg/kg;16% by volume) consumption
Population: as for outcome 5
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Placebo | Carisbamate
Number analyzed (Participants) | 8 | 8
beats per minute
  'Pulse' + 15 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 81.8 (4.0) | 86.5 (5.3)
  'Pulse' + 30 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 83.3 (2.0) | 90.1 (4.8)
  'Pulse' + 60 minutes after alcohol (0.8g/kg; 16% by volume) consumption | 81.8 (2.5) | 91.0 (5.5)

ADVERSE EVENTS:
Time Frame: Adverse event data was assessed over the 4 week active enrollment period on each condition (active carisbamate vs. placebo), up to 8 weeks following active enrollment.
Groups:
- Placebo First, Then Carisbamate: Participants will receive placebo from days 2- 4.
  Placebo: Placebo treatment only
- Carisbamate First, Then Placebo: Participants will receive carisbamate 600mg qd from days 2- 4.
  Carisbamate: 600mg Orally on days 2-4
Arm/Group | Placebo First, Then Carisbamate | Carisbamate First, Then Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall have the right to publish or otherwise publicly disclose information gained in the course of this Agreement. Investigator agrees to submit to Company copies of manuscripts, posters, slides, or abstracts that are intended for presentation or publication and that contain the results of the performance of this Agreement not less than 30 days before submission of manuscripts for publications or presentations of slides and posters, or 10 days prior to abstract submission.

DOCUMENTS (1):
  • Informed Consent Form (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT02435381/ICF_000.pdf